CLINICAL TRIAL: NCT02429830
Title: A Prospective, Multicenter Study of REflux Management With the LINX® System for Gastroesophageal REFlux Disease After Laparoscopic Sleeve Gastrectomy
Brief Title: LINX Reflux Management System in Subjects With GERD Who Have Previously Undergone a Laparoscopic Sleeve Gastrectomy
Acronym: RELIEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Torax Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4600; TRX_2016_01 (Other: Ethicon Endosurgery (Industry Sponsor))
Record Dates: First submitted 2015-04-13; First posted 2015-04-29 (Estimated); Results first posted 2022-07-05 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: GERD; Gastroesophageal Reflux Disease
Keywords: gastroesophageal reflux disease; GERD; obesity; LSG; Laparoscopic Sleeve Gastrectomy
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single arm study (Other): Previous LSG patient will be treated with the LINX device and serve as their own control
  Interventions: Device: LINX device

INTERVENTIONS:
Device: LINX device — The LINX device is a permanent implant placed at the area of the lower esophageal sphincter (LES) and is designed to augment a weak LES and minimize or eliminate GERD-related symptoms.

SUMMARY:
The purpose of this study is to evaluate the LINX device in patients who have previously undergone laparoscopic sleeve gastrectomy (LSG) for obesity and have chronic gastroesophageal reflux disease (GERD). The study will monitor safety and changes in reflux symptoms.

DETAILED DESCRIPTION:
The objective of this study is to confirm safety and efficacy after laparoscopic sleeve gastrectomy (LSG) in subjects indicated for LINX is similar to the outcomes that formed the basis for the LINX Premarket Approval to support modification of the current labeling. Presently, there is a precautionary statement that safety and effectiveness of the LINX has not been established for prior esophageal or gastric surgery or endoscopic intervention.

Patients with GERD that have undergone a LSG procedure have limited surgical treatment options if they are looking for an alternative to continuous acid suppression therapy (i.e. proton pump inhibitors or equivalent). One procedure, fundoplication, is extremely difficult to perform as LSG patients have a limited amount of fundus tissue remaining after sleeve surgery. Roux-en-Y gastric bypass (RYGB) may be chosen as a conversion procedure but is more invasive with the potential for serious complications. LINX may be considered as an alternative and less invasive option that may potentially have few complications compared to RYGB.

The study is an observational, multicenter, single-arm study with prospective enrollment. Based on the observational status of the study, no formal statistical hypothesis tests will be conducted. Up to 30 patients meeting the eligibility requirements will be implanted with LINX and followed through 12-months after implant. Up to twelve (12) clinical sites will enroll subjects. Safety evaluations will be ongoing throughout the duration of the study, starting at the implant procedure. Efficacy endpoints will be evaluated at the 12-month visit.

Safety will be evaluated based on the rate of serious device and procedure related adverse events (AEs). Safety will also be evaluated by endoscopy to assess the mucosa and x-rays to verify device location at 12 months post implant. Efficacy will be measured at 12 months (compared to baseline) by examining 3 variables: normalization of total distal acid exposure or at least a 50% reduction, at least a 50% reduction in total GERD-HRQL scores and at least a 50% reduction in average daily PPI dosage.

ELIGIBILITY:
INCLUSION CRITERIA

Subjects included in the study must meet all the following criteria:

1. Age >22 years
2. Laparoscopic sleeve gastrectomy (LSG) for obesity >12 months prior to proposed device implantation date.
3. Subject is a surgical candidate, i.e. is able to undergo general anesthesia and laparoscopic surgery.
4. Documented typical symptoms of GERD for longer than 6 months (regurgitation or heartburn which is defined as a burning epigastric or substernal pain which responds to acid neutralization or suppression).
5. Subject requires daily proton pump inhibitor or other anti-reflux drug therapy.
6. Total distal ambulatory esophageal pH must meet the following criteria: pH <4 for >4.5% of the time. Note: Subjects shall have discontinued any GERD medications for at least 7 days prior to testing, with the exception of antacids up to the morning of testing.
7. Subjects with symptomatic improvement on PPI therapy demonstrated by a GERD-HRQL score of <10 on PPI and >15 off PPI, or subjects with a >6 point improvement when comparing their on PPI and off PPI GERD-HRQL scores.
8. GERD symptoms, in absence of PPI therapy (minimum 7 days).
9. If the subject is of child bearing potential must have a negative pregnancy test within one week prior to implant and must agree to use effective means of birth control during the course of the study.
10. Subject is willing and able to cooperate with follow-up examinations
11. Subject has been informed of the study procedures and the treatment and has signed an informed consent form.

EXCLUSION CRITERIA

Subjects should be excluded from the study based on the following criteria:

1. The procedure is an emergency procedure.
2. Suspected or known allergies to titanium, stainless steel, nickel, or ferrous materials.
3. Presence of ˃3 cm hiatal hernia as determined by endoscopy or barium esophagram.
4. Subject had any major complications related to the laparoscopic sleeve gastrectomy that may interfere with, or increase the risks of the LINX procedure (such as, but not limited to, leaks from the gastric remnant and infection at the sleeve gastrectomy)
5. Plans to surgically revise the gastric pouch (either known preoperatively or decided intraoperatively)
6. Currently being treated with another investigational drug or investigational device.
7. Suspected or confirmed esophageal or gastric cancer or prior gastric or esophageal surgery or endoscopic intervention for GERD (with the exception of sleeve gastrectomy).
8. Distal amplitude <35 mmHg or <70% peristaltic sequences (if using Conventional Manometry). -or- If using High Resolution Manometry (exclude for any of the following):

   * Distal Contractile Integral (DCI) ≤ 450 mmHg·s·cm or
   * ≥ 50% ineffective swallows or
   * ≥ 50% fragmented swallows (Fragmented swallows are defined as those with a ≥ 5cm break [large] in peristaltic integrity).
9. Presence of esophagitis - Grade C or D (LA Classification).
10. BMI >35.
11. Symptoms of dysphagia more than once per week within the last 3 months.
12. Diagnosed with Scleroderma.
13. Diagnosed with an esophageal motility disorder such as but not limited to achalasia, nutcracker esophagus, or diffuse esophageal spasm or hypertensive LES.
14. Subject has a history of or known esophageal stricture or gross esophageal anatomic abnormalities (Schatzki's ring, obstructive lesions, etc.)
15. Subject has esophageal or gastric varices
16. History of/or known Barrett's esophagus. Note: The diagnosis of Barrett's esophagus requires both endoscopic and histologic evidence of metaplastic columnar epithelium. Endoscopically, there must be columnar epithelium within the esophagus. Histologically, the epithelium must be metaplastic, as defined by the presence of goblet cells.by
17. Subject cannot understand trial requirements or is unable to comply with follow-up schedule
18. Pregnant or nursing, or plans to become pregnant during the course of the study.
19. Any reason which the Investigator believes may cause the subject to be non-compliant with or unable to meet the protocol requirements.
20. Subject has an electrical implant or metallic, abdominal implants.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Petraiuolo, MD, Study Director — Ethicon Endo-Surgery
Locations (12):
- United States (12):
  - Northwest Allied Bariatric & Foregut Surgery, Tucson, Arizona
  - Mercy Health Northwest Arkansas, Rogers, Arkansas
  - Keck Medical Center of USC, Los Angeles, California
  - Institute of Esophageal and Reflux Surgery, Englewood, Colorado
  - RWJBH Univ. Hospital Somerset/Advanced Surgical and Bariatrics of NJ, PA, Somerset, New Jersey
  - Buffalo General Medical Center, Buffalo, New York
  - Adirondack Surgical Group, Saranac Lake, New York
  - East Carolina University, Greenville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Coastal Carolina Bariatric & Surgical Center, Summerville, South Carolina
  - Panhandle Weight Loss Center, Amarillo, Texas
  - Gunderson Health System, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LINX Device: Participants with gastroesophageal reflux disease (GERD) who previously underwent a laparoscopic sleeve gastrectomy were treated with the LINX Reflux Management System, a laparoscopic, fundic-sparing anti-reflux device designed to augment a weak lower esophageal sphincter (LES) and minimize or eliminate GERD-related symptoms.
Period: Overall Study
Arm/Group | LINX Device
Started | 30
Completed | 27
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Device Explant | 2

BASELINE CHARACTERISTICS:
Arm/Group | LINX Device
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Greater Than or Equal to (>=) 50 Percent (%) Reduction in Total Gastroesophageal Reflux Disease (GERD)- Health-Related Quality of Life (HRQL) Score Compared to Baseline (Off GERD Medications) at the 12-month Follow-up
Description: Percentage of participants reporting >=50% reduction in total GERD-HRQL score compared to baseline (off GERD Medications) at the 12-month follow-up were reported. The GERD-HRQL score consisted of 10 questions, where participants were required to answer each question on a scale of 0 to 5 (0: no symptoms; 1: symptoms noticeable but not bothersome; 2: symptoms noticeable and bothersome but not every day; 3: symptoms bothersome every day; 4: symptoms affect daily activity; 5: symptoms are incapacitating, unable to do activities). The total score was derived by simply adding the individual score of each question. The total score ranged from 0 to 50 where a higher score indicated more severe disease. The best possible total GERD-HRQL score was 0 (asymptomatic in all questions) and the worst possible score was 50 (incapacitated in all questions).
Time Frame: Up to 12 Months
Population: The Full Analysis Set (FAS) consisted of participants who met all eligibility criteria, provided informed consent, completed baseline assessments, and underwent a LINX procedure. Here, 'N' (Number of participants analyzed) included all participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | LINX Device
Number analyzed (Participants) | 26
Percentage of participants | 80.8

2. Primary Outcome: Percentage of Participants Reporting Normalization of Total Distal Acid Exposure Time or at Least a 50% Reduction in Total Distal Acid Exposure Time Compared to Baseline at the 12-month Follow-up
Description: Percentage of participants reporting normalization of total distal acid exposure time or at least a 50% reduction in total distal acid at the 12-month follow-up were reported. The testing was performed by a reflux sensing implantable capsule (for example, Bravo) or via a trans-nasal catheter. Success of the LINX device in decreasing abnormal levels of gastric acid in the esophagus was defined as normalization of distal acid exposure time (pH less than [<] 4 for greater than or equal to [>=] 4.5% of monitoring time) or at least 50% reduction in distal acid exposure time compared to baseline.
Time Frame: Up to 12 months
Population: The FAS consisted of participants who met all eligibility criteria, provided informed consent, completed baseline assessments, and underwent a LINX procedure. Here, 'N' (Number of participants analyzed) included all participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | LINX Device
Number analyzed (Participants) | 27
Percentage of participants | 44.4

3. Primary Outcome: Percentage of Participants Reporting >=50% Reduction in Average Daily Protocol Pump Inhibitors (PPIs) Dosage Compared to Baseline at the 12-month Follow-up
Description: Percentage of participants reporting >=50% reduction in average daily protocol pump inhibitors (PPIs) dosage compared to baseline at the 12-month follow-up were reported.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | LINX Device
Number analyzed (Participants) | 24
Percentage of participants | 95.8

4. Primary Outcome: Number of Participants Experiencing Serious Device and/or Procedure Related Adverse Events After LINX Placement Out to 12 Months
Description: Number of participants experiencing serious device and/or procedure related adverse events after LINX placement out to 12 months were reported. SAE is any AE that results in: requires subject hospitalization greater than (>) 24 hours; is life-threatening or results in death; requires prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; results in fetal distress, fetal death, or a congenital anomaly or birth defect; requires intervention to prevent permanent impairment or damage of body function or structure; other serious important medical events that do not fit in the other outcomes and may jeopardize the participant and may require medical or surgical intervention to prevent one of the other outcomes.
Time Frame: Up to 12 months
Population: The FAS consisted of participants who met all eligibility criteria, provided informed consent, completed baseline assessments, and underwent a LINX procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | LINX Device
Number analyzed (Participants) | 30
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Full Analysis Set (FAS) consisted of participants who met all eligibility criteria, provided informed consent, completed baseline assessments, and underwent a LINX procedure.
Arm/Group | LINX Device
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 15/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LINX Device (N=30)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Pain (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LINX Device (N=30)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Pain (Surgical and medical procedures) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Esophageal spasm (Gastrointestinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epigastric pain and bloating (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Face tingling and pain (Skin and subcutaneous tissue disorders) | 1 (1)
Foam pooling in throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypersensitivity to Dermabond (Skin and subcutaneous tissue disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post-Op Atelectasis & pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting, pain in chest and nausea (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the complete nor any part of the results of the study carried out under this protocol, nor any of the information provided by the Sponsor for the purposes of performing the study, will be published or passed on to any third party without the written consent of Sponsor. Any Investigator involved with this study is obligated to provide the Sponsor with complete test results and all data derived from the study.

DOCUMENTS (2):
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT02429830/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT02429830/SAP_001.pdf